CLINICAL TRIAL: NCT00305279
Title: The Effects of Dietary Phosphate Intake on Calciotropic Hormones and FGF23
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: H40550-27771; 1K23RR020343 (NIH)
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Healthy; Kidney Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Diet

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- 1 (Active Comparator)
  Interventions: Other: Dietary
- 2 (Active Comparator)
  Interventions: Other: Dietary
- 3 (Active Comparator)
  Interventions: Other: Dietary

INTERVENTIONS:
Other: Dietary — Dietary
  Arms: 1
Other: Dietary — Dietary
  Arms: 2
Other: Dietary — Dietary
  Arms: 3

SUMMARY:
The purpose of this study is to determine the effects of different amounts of phosphorus in the diet on hormones that control phosphorus and bone health both in people who are healthy and in ones who have moderate kidney disease.

DETAILED DESCRIPTION:
Chronic kidney disease affects 11% of the US population; over half of those affected have skeletal manifestations of their renal disease. Renal osteodystrophy is a complex disease, in which multiple mineral systems and related hormones play a role, including phosphate homeostasis. Phosphate regulation primarily depends on renal handling of phosphate, which is partly controlled by parathyroid hormone and vitamin D. However, other mediators in this system clearly exist. Recently, evidence has been accruing that one such factor may be FGF23, a protein produced by osteogenic cells. States of excess FGF23 are associated with marked phosphate wasting, hypophosphatemia, osteomalacia, and inappropriately low calcitriol. FGF23 levels are measurable in healthy humans and markedly elevated in patients who require hemodialysis, although its physiologic role in either state is unknown. Some retrospective evidence suggests that FGF23 is affected by phosphate intake. We are performing a study to gather data describing the response of FGF23 to changes in dietary phosphorus intake in healthy men and women and in men and women with moderate renal insufficiency. The specific aims of this pilot study are: 1) To examine the physiologic effects of alterations in dietary phosphorus on FGF23 in healthy subjects; 2) To examine the physiologic response of FGF23 to dietary phosphorus alterations in patients with moderate renal failure; and 3) To assess whether serum levels of 1,25-dihydroxyvitamin D vary inversely with those of FGF23 when dietary phosphate is changed. The proposed research plan is a dietary intervention trial in which we will study the response of serum FGF23 levels to diets with varying phosphorus contents in healthy adults and adults with moderate renal insufficiency.

ELIGIBILITY:
Inclusion Criteria:

HEALTHY SUBJECTS:

* Men 21-65 years of age;
* Premenopausal women over 21 years of age taking oral contraceptives;
* Postmenopausal women less than 65 years of age;

CHRONIC KIDNEY DISEASE SUBJECTS:

* Men 21-65 years of age;
* Premenopausal women over 21 years of age taking oral contraceptives;
* Postmenopausal women less than 65 years of age;
* Creatinine clearance between 30 and 59 ml/min/1.73 m2 as calculated using the equation derived from the Modification of Diet in Renal Disease (MDRD) study.

Exclusion Criteria:

* Medications affecting bone metabolism;
* Abnormal liver or GI function;
* Extreme electrolyte abnormalities;
* BMI >30 kg/m2.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-02; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Hormonal regulators of mineral metabolism | Last two days of each intervention phase

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Antoniucci, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States